CLINICAL TRIAL: NCT03209219
Title: Randomized Prospective Comparative Study of Interferon α2a and Cyclosporine in Patients With Refractory Behçet's Disease Uveitis
Brief Title: Interferon α2a Versus Cyclosporine for Refractory Behçet's Disease Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Meifen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z171100001017217
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Behçet Disease; Uveitis
Keywords: effectiveness, safety
MeSH Terms: conditions — Behcet Syndrome; Uveitis | interventions — Interferon alpha-2; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferon Alpha 2A (Experimental): Patients are treated with IFNα2a 3×10^IU α2a by subcutaneous injection or intramuscular injection daily for 4 weeks, and followed by every other day there after.
  Interventions: Drug: Interferon Alfa-2A
- Cyclosporine (Active Comparator): Patients are treated with oral CsA 100mg twice daily.
  Interventions: Drug: Cyclosporine Pill

INTERVENTIONS:
Drug: Interferon Alfa-2A — 3×10^6 IU， subcutaneous or intramuscular injection, qd for × 4 weeks, and qod thereafter
  Arms: Interferon Alpha 2A
Drug: Cyclosporine Pill — 100mg， oral, bid
  Arms: Cyclosporine

SUMMARY:
Brief summary: This study compares the long-term efficacy and safety of interferon (IFN) α2a and cyclosporine (cyclosporin A, CsA) following suppression of acute attack by high-dose oral glucocorticosteroid in patients with refractory Behçet's uveitis (BDU). Half of the participants will receive IFNα2a while the other half will receive CsA.

DETAILED DESCRIPTION:
Detailed description: Both CsA and IFNα2a have been shown to be effective for long-term control of BDU, however, randomized prospective comparative studies are scarce, particularly in East Asian populations. Our preliminary data gave us the impression that IFNα2a might be more effectiveness than CsA in long-term control of refractory BDU, and this study aimed to compare their effectiveness and safety profiles in a well-designed prospective study. Refractory BDU is defined as relapse of posterior or pan- uveitis with at least 10mg daily prednisone (or equivalent) and one traditional immunomodulatory treatment (IMT) agents. The acute attack is controlled with large dose oral corticosteroid (60mg daily prednisone) for 4 weeks, and then the patients are randomly assigned to the IFN arm and the CsA arm, in which patients are treated with IFNα2a (3×10^6 IU qd for 4 weeks and qod thereafter) and CsA (100mg bid), respectively, along with a fixed tapering regimen of corticosteroid. Patients were followed up until relapse, or for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Refractory BDU patients fulfilling the International Criteria for Behçet's disease (ICBD) published in 2013 with recent recurrence of pan- or posterior uveitis;
* The patient should be on ≥10mg/d oral prednisone or equivalent with at least one of the following IMT agents: cyclophosphamide≥50mg/d, CsA≥100mg/d, azathioprine≥50mg/d, methotrexate≥15mg/w, mycophenolate≥1000mg/d, tacrolimus≥2mg/d.

Exclusion Criteria:

* Previous treatment with interferon-α;
* Pregnancy, breast feeding women;
* Malignancy;
* Renal impairment (creatinine > 1.5 mg/dl);
* Uncontrolled hypertension or diabetes;
* Depression or other psychic disorders;
* History of acute or chronic inflammatory joint or autoimmune disease;
* Patients with severe extra-ocular involvement other than oral/genital ulcer and skin involvement;
* Organ or bone marrow transplant recipient, cardiac failure > NYHA III;
* Acute liver disease with ALT or SGPT 2x above normal;
* White blood cell count < 3500/mm^3;
* Platelet count < 100000/mm^3;
* Hgb < 8.5g/dl;
* T-SPOT TB: ≥200 SFCs per 10^6 PBMC;
* Active peptic ulcer, systemic or local infection, moderate to severe osteoporosis or other contraindications of large dose corticosteroids;
* Previous intolerance to CsA;
* Other severe ocular diseases or intraocular surgery within 3 months;
* Media opacity precluding a clear view of the fundus;
* Positive screen test for HBV, HCV, HIV infection or syphilis;
* Body weight <45 kg;
* Alcohol abuse or drug abuse;
* Mental impairment;
* Uncooperative attitude.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Response rate | Within the 12-month follow-up period
  Percentage of participants who achieve complete remission or partial remission
Complete remission rate | Within the 12-month follow-up period
  Percentage of participants who achieve complete remission without relapse of posterior or pan-uveitis
Tolerance rate | Within the 12-month follow-up period
  Percentage of participants who adhere to the treatment without severe side effects

SECONDARY OUTCOMES:
Time to reach complete remission | Within the 12-month follow-up period
  The time from the therapy initiation to a complete absence of ocular inflammation for complete responders
Duration of relapse-free | within the 12-month follow-up period
  The duration between the therapy initiation to the relapse for partial responders and nonresponders
BCVA | Within the 12-month follow-up period
  Changes of best-corrected visual acuity
BOS24 score | Within the 12-month follow-up period
  Score of ocular inflammation using the Behcet disease ocular attack score 24 (BOS24)
Glucocorticoid-sparing effect | Within the 12-month follow-up period
  Changes of corticosteroid dosage
Incidence of adverse effects | Within the 12-month follow-up period
  Incidence of adverse effects
Incidence of significant abnormal changes in vital signs or laboratory test results | Within the 12-month follow-up period
  Incidence of significant abnormal changes in vital signs or laboratory test results
Adverse effects profile | Within the 12-month follow-up period
  Types of drug adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data are available from the investigator upon reasonable request.